CLINICAL TRIAL: NCT02835508
Title: A Single-Dose, Open-Label, Randomized, Parallel-Group Study to Assess the Pharmacokinetic Profile of JNJ-56021927 When Administered as the Tablet Formulation in Healthy Male Japanese Subjects
Brief Title: Pharmacokinetic Study of JNJ-56021927 When Taken Orally as Tablet Formulation in Healthy Male Japanese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108165; 56021927PCR1021 (Other: Janssen Pharmaceutical K.K.)
Record Dates: First submitted 2016-06-29; First posted 2016-07-18 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Healthy
MeSH Terms: interventions — apalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Experimental): Participants will receive a single dose of 1 tablet of JNJ-56021927, 60 milligram (mg) on Day 1.
  Interventions: Drug: JNJ-56021927 60 Milligram
- Treatment B (Experimental): Participants will receive a single dose of JNJ-56021927, 120 mg (2 tablets*60 mg) on Day 1.
  Interventions: Drug: JNJ-56021927 120 Milligram
- Treatment C (Experimental): Participants will receive a single dose of JNJ-56021927, 240 mg (4 tablets*60 mg) on Day 1.
  Interventions: Drug: JNJ-56021927 240 Milligram

INTERVENTIONS:
Drug: JNJ-56021927 60 Milligram — JNJ-56021927 60 mg oral tablet.
  Other Names: apalutamide
  Arms: Treatment A
Drug: JNJ-56021927 120 Milligram — JNJ-56021927 120 mg as 2 tablets of 60 mg.
  Other Names: apalutamide
  Arms: Treatment B
Drug: JNJ-56021927 240 Milligram — JNJ-56021927 240 mg as 4 tablets of 60 mg.
  Other Names: apalutamide
  Arms: Treatment C

SUMMARY:
The purpose of the study is to assess the safety and Pharmacokinetic (PK) profile of JNJ-56021927 and its active metabolite JNJ-56142060 after single-dose administration of 60 milligram (mg), 120 mg, and 240 mg JNJ-56021927 as the tablet formulation in healthy male Japanese participants.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have a body mass index between 18.0 and 29.9 Kilogram per meter square (kg/m^2), inclusive, and a body weight not less than 50 Kilogram (kg)
* Participant must have a blood pressure between 90 and 140 Millimeters of Mercury (mm Hg) systolic, inclusive, and no higher than 90 mm Hg diastolic at screening
* Participant must have a normal 12-lead Electrocardiogram (ECG) (based on the mean value of the triplicate parameters) consistent with normal cardiac conduction and function at screening, including: a) normal sinus rhythm (heart rate between 45 and 90 beats per minute, extremes included); b) QT interval corrected for heart rate according to Fridericia (QTcF) <= 450 milliseconds (ms); c) QRS interval less than or equal (<=)110 ms; d) PR interval <200 ms; e) ECG morphology consistent with healthy cardiac conduction and function
* Participant must be a healthy Japanese male
* Participant must agree to use an adequate contraception method as deemed appropriate by the investigator; to always use a condom during intercourse and to not donate sperm during the study and for 3 months after study drug administration

Exclusion Criteria:

* Participant with a history of current clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, hepatic or renal insufficiency, thyroid disease, neurologic or psychiatric disease, infection, or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Participant has donated blood or blood product or had substantial loss of blood more than 200 milliliter (mL) within 1 month before study drug administration, or greater than equal (>=) 400 mL within 3 months before study drug administration, or participant has donated a total volume of blood in the past one year exceeding 1200 mL, or participant has an intention to donate blood or blood products during the study and for at least 2 months after completion of the study
* Participant has presence of sexual dysfunction (abnormal libido, erectile dysfunction, etc) or any medical condition that would affect sexual function
* Participant has received an investigational drug including investigational vaccines or used an invasive investigational medical device within 3 months or within a period less than 10 times the drug's half-life, whichever is longer, before the planned study drug administration
* Participant has a history of hepatitis B surface antigen (HBsAg) or hepatitis C antibody (anti-hepatitis C virus {HCV}) positive, or other clinically active liver disease, or tests positive for HBsAg or anti-HCV at screening

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2016-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | Predose, Up to Day 57
  Maximum observed plasma concentration (Cmax) will be assessed.
Time to Reach Maximum Observed Plasma Concentration (Tmax) | Predose, Up to Day 57
  Actual sampling time to reach maximum observed analyte concentration (Tmax) will be assessed.
Area Under Concentration from time zero to the last quantifiable AUC (0-last) | Predose, Up to Day 57
  AUC from time zero to the last quantifiable concentration will be assessed.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) | Predose, Up to Day 57
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC (0-last) and C (0-last)/lambda(z); wherein AUC (0-last) is area under the plasma concentration-time curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda (z) is elimination rate constant. AUC (0-infinity) will be assessed.
Time to Last Quantifiable Plasma Concentration (Tlast) | Predose, Up to Day 57
  The Tlast, time to last observed quantifiable plasma concentration will be assessed.
Percentage of Area Under the Plasma Concentration-Time Curve Extrapolated From Last Measurable Concentration to Infinite Time (%AUC,ext) | Predose, Up to Day 57
  Percentage of area under the plasma concentration-time curve extrapolated from last measurable concentration to infinite time (%AUC,ext) is calculated as (AUC [0-infinity] minus AUC [0-last])/ AUC [0-infinity])*100.
Apparent Clearance (CL/F) | Predose, Up to Day 57
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood. CL/F will be calculated as CL/F = Dose/AUC [0-infinity]
Apparent Terminal Elimination Half-life (t1/2term) | Predose, Up to Day 57
  Apparent terminal elimination half-life, calculated as 0.693/apparent terminal elimination rate constant (λz)
Apparent Terminal Elimination Rate Constant (lambda z) | Predose, Up to Day 57
  Apparent terminal elimination rate constant, estimated by linear regression using the terminal log-linear phase of the log transformed concentration vs time data
Apparent Volume of Distribution (Vd/F) | Predose, Up to Day 57
  Apparent volume of distribution based on the terminal phase following oral administration calculated as Vd/F = Dose/ apparent terminal elimination rate constant (λz)*AUC [0-infinity]
Metabolite to Parent Drug Ratio for Maximum Observed Plasma Concentration (MPR Cmax) | Predose, Up to Day 57
  Metabolite to parent drug ratio for Cmax will be assessed.
Metabolite to Parent Drug Ratio for Area Under Concentration from time zero to the last quantifiable concentration (MPR AUC [0-last]) | Predose, Up to Day 57
  Metabolite to parent drug ratio for AUC [0-last] will be assessed.
Metabolite to Parent Drug Ratio for Area Under Curve from time zero extrapolated to infinity (MPR AUC [0-infinity]) | Predose, Up to Day 57
  Metabolite to parent drug ratio for AUC [0-infinity] will be assessed.
Area Under Curve from time of administration to 24 hours post dosing | Predose, Up to Day 57
  AUC from time of administration to 24 hours post dosing will be assessed.
Area Under Curve from time of administration to 168 hours post dosing | Predose, Up to Day 57
  AUC from time of administration to 168 hours post dosing will be assessed.

SECONDARY OUTCOMES:
Number of Participants With Adverse Events as a Measure of Safety and Tolerability | Up to Day 57

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K. Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (1):
- Kumamoto, Japan